CLINICAL TRIAL: NCT05112575
Title: Evaluation of Patient Stress Level Caused by Radiological Investigations in Early Postoperative Phase After Craniotomy (IPAST-CRANIO): Protocol of a Swiss Prospective Cohort Study
Brief Title: Evaluation of Patient Stress Level Caused by Radiological Investigations in Early Postoperative Phase After Craniotomy
Acronym: IPAST-CRANIO
Status: Terminated | Type: Observational
Why Stopped: Failed resources.
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-01590
Record Dates: First submitted 2021-09-16; First posted 2021-11-09 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Pain; Postoperative Nausea
Keywords: Magnetic resonance imaging; Craniotomy; Postoperative imaging
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early imaging: within 36 hours postoperatively.: Patients fulfilling eligibility criteria between 18 and 80 years old who receive MRI or CT follow-up after craniotomy for resection of a space occupying lesion (benign or malignant) or vascular within 36 hours after neurosurgical procedure.
  Interventions: Radiation: Postoperative imaging with magnetic resonance imaging or computed tomography
- Late imaging: between 36 and 72 hours postoperatively: Patients fulfilling eligibility criteria between 18 and 80 years old who receive MRI or CT follow-up after craniotomy for resection of a space occupying lesion (benign or malignant) or vascular between 36 and 72 hours after neurosurgical procedure.
  Interventions: Radiation: Postoperative imaging with magnetic resonance imaging or computed tomography

INTERVENTIONS:
Radiation: Postoperative imaging with magnetic resonance imaging or computed tomography — Postoperative imaging control with magnetic resonance or computed tomography after craniotomy for vascular or neurooncological operations.

SUMMARY:
Postoperative imaging after neurosurgical intervention is usually performed in the first 72 hours after surgery. Postoperative radiological examinations in the first 72 hours provide accurate assessment of postoperative resection status. On the other side is frequently reported by patients that the earlier postoperative examinations after craniotomy for tumor and vascular procedures are associated with distress, exertion, nausea, and pain. Therefore, psychological and physical stress on the patient could be a potential disadvantage of earlier (up to 36 hours postoperatively) follow-up. The goal of this study is to evaluate and determine the optimal time frame for postoperative imaging with MRI and CT in terms of medical and neuroradiological implications and patient's subjective stress.

The primary endpoint of the study is the extent of subjective distress due to postoperative MRI and CT monitoring in relation to the time interval after surgery Data will be prospectively collected from all patients aged 18 to 80 years who receive postoperative MRI or CT follow-up after craniotomy for resection of a cerebral tumor (benign and malignant) or vascular surgery.

This study determines, whether a timing of postoperative imaging can improve patient satisfaction and reduce pain, stress and discomfort caused by postoperative imaging. The outcome corresponds to the value-based medicine approach of modern patient-centred medicine. Results will be published in peer-reviewed journals and electronic patient data will be safely stored for 15 years.

DETAILED DESCRIPTION:
Background and rationale Magnetic resonance imaging (MRI) after neurosurgical resection of a cerebral tumor is usually performed in the first 72 hours after surgery. 1-4 Accurate assessment of early postoperative resection status in brain tumors is mandatory for further treatment planning, e.g., delineation of the radiation field in radiotherapy, or reoperation for significant residual tumor. 5 Various MRI-sequences provide information on tumor size and location, as well as additional insight into secondary phenomena such as edema, hemorrhage, infarct, necrosis, and signs of increased intracranial pressure. 1, 3, 5, 6 The 72 hours' time window is crucial for accurate assessment of resection status and is additionally used for quality control of the neurosurgical procedure. 7 Postoperative MRI later than 72 hours after surgery can lead to false positive contrast enhancement due to absorption of contrast in the surgical area which can complicate the assessment of resection status. 1, 6 Postsurgical repair mechanisms at the resection site that result from hypervascularization and disruption of blood-brain barrier are probably responsible for this delayed enhancement. 7 The potential advantages of early imaging (within 36 hours after surgery) are better radiological assessment of the surgical site and earlier diagnosis of postoperative complications, such as infarcts, postoperative bleeding or edema. This may help in improving the postoperative management of patients with complications. Moreover, earlier information about the outcome of surgery could also lead to psychological relief for patients in the early postoperative period. Disadvantages of early postoperative examinations after craniotomy are frequently reported by patients and include distress, exertion, nausea, and pain during and after the examination. As such, psychological and physical patient stress could be a potential disadvantage of early (within 36 hours after surgery) MRI examination. An alternative image modality is Computed Tomography (CT), which may be less stressful for the patients because it takes only 5 to 10 minutes to complete the scan and the patients do not have to lie in small claustrophobic space compared to MRI. However, with this modality the postoperative resection status cannot reliably be assessed. To the authors knowledge, no previous literature has been published which addressed the stress factors during postoperative imaging. To authors opinion, a more patient-centered view regarding postoperative MRI investigation needs more clarification, so the authors want to investigate the intensity of patient stress after postoperative imaging at different intervals from surgery. With optimization of the time window of the MRI examination, the authors want to improve the psychological and physical patient stress, which may have a positive influence on early recovery. Additionally, establishing an optimal time window for postoperative MRI imaging will help in scheduling the examination before the elective surgical treatment. This will have a positive impact on preparing patients, radiology employees, nurses and physicians for a smooth and easy transport to and from the MRI examination.

Objectives The goal of this study is to assess whether early imaging with MRI (within 36 hours) after craniotomy is different regarding patient stress, than delayed imaging (between 36 and 72 hours). Secondly, the authors want to assess whether there is a difference in patient stress level between postoperative MRI and CT within 72 hours postoperatively.

The authors hypothesize that delayed imaging with MRI after craniotomy is more comfortable for patients without negative implication of radiological assessment, than imaging within 36 hours. Secondly, the authors hypothesize that postoperative MRI is more stressful for patients than CT.

Trial design The IPAST-CRANIO study (Evaluation of patient STress level caused by radiological Investigations in early Postoperative phase After CRANIOtomy) is a patient-oriented, prospective, exploratory cohort study.

Methods: Participants, interventions and outcomes Data will be collected from patients between 18 and 80 years old who receive MRI or CT follow-up after craniotomy for resection of a space occupying lesion (benign or malignant) or vascular procedure at the Department of Neurosurgery at the University Hospital Zurich

ELIGIBILITY:
Inclusion Criteria:

* Written consent of the patient
* Age between 18 and 80 years
* Planned for supra- or infratentorial (partial) resection of space occupying lesion (benign or malignant) or vascular neurosurgical procedure (clipping of an aneurysm, resection of an arteriovenous malformation, resection of cavernoma)
* Patients planned for MRI or CT follow-up within 72 hours after surgery

Exclusion Criteria:

* No informed consent
* Operation using only one burr hole (e.g. biopsy)
* Not able to fill out the questionnaires due to cognitive impairment or aphasia
* Not understanding German or English language
* Contraindication for MRI examination
* No postoperative MRI or CT examination planned within 72 hours after surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be collected from patients between 18 and 80 years old who receive MRI or CT follow-up after craniotomy for resection of a space occupying lesion (benign or malignant) or for any vascular procedure at the Department of Neurosurgery at the University Hospital Zurich
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is the difference in subjective distress after craniotomy, measured just before and after postoperative MRI or CT. | The measurements are taken up to 1 hour before and up to 1 hour after postoperative radiological imaging after craniotomy.
  Subjective distress is evaluated as a combination of the results of the 3 scores: visual analogue scale for (VAS) pain, VAS for nausea and Body Part Discomfort score.

SECONDARY OUTCOMES:
Patient specific secondary endpoint | The measurement is taken up to 1 hour after postoperative radiological imaging after craniotomy.
  Patient subjective interpretation of whether MRI control was performed at the correct interval. At the end of the questionnaire, patients will be asked to answer the following question:
  In your opinion, should the MRI and/or CT scan have been performed earlier or later? The possible answers are:
  * Yes, earlier;
  * Yes, later;
  * No, I am satisfied with the timing of the exam.
Radiology specific secondary endpoints | The radiological evaluation of imaging after craniotomy is performed up to 12 hours after postoperative radiological examination.
  Presence of residual tumor on MRI: yes or no. Presence of contrast enhancement on MRI (postoperative reactive change, not tumor specific): yes or no.
  Presence of post-operative bleeding on CT or MRI: yes or no. Presence of postop-operative infarction on MRI: yes or no Residual perfusion of the aneurysm or AVM remnant on MRI or CT: yes or no.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Tosic L, Thoma M, Voglis S, Hofer AS, Bektas D, Pangalu A, Regli L, Germans MR. Evaluation of patient STress level caused by radiological Investigations in early Postoperative phase After CRANIOtomy (IPAST-CRANIO): protocol of a Swiss prospective cohort study. BMJ Open. 2022 Sep 21;12(9):e061452. doi: 10.1136/bmjopen-2022-061452. PMID 36130762